CLINICAL TRIAL: NCT00847262
Title: Hypertension With Obesity Trial: Diabetes Mellitus Branch
Brief Title: Trial Comparing Metabolic Effects of Telmisartan and Amlodipine on Hypertensive Patients With Obesity and Diabetes
Acronym: HOT-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Chief of the Department of Hypertension & Endocrinology, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOT-2
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension; Obesity; Diabetes
Keywords: Hypertension; Abdominal obesity; Diabetes; Treatment
MeSH Terms: conditions — Hypertension; Obesity; Diabetes Mellitus; Obesity, Abdominal | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telmisartan Group (Experimental): Telmisartan intervention group
  Interventions: Drug: Temisartan
- Amlodipine Group (Active Comparator): Amlodipine intervention group
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Temisartan — Temisartan, initial dose: 40 mg per day, Max dose: 160 mg per day
  Arms: Telmisartan Group
Drug: Amlodipine — Amlodipine, initial dose: 5 mg per day, Max dose: 10 mg per day
  Arms: Amlodipine Group

SUMMARY:
Recent studies have shown that obese people are more prone to high blood pressure. With the co-existence of obesity, hypertension and diabetes, patients were more susceptible to hyperlipidemia, coronary and cerebral atherosclerosis and peripheral vascular disease. Abdominal obesity has often accompanied by substantial accumulation of visceral fat, which increased secretion of many inflammatory mediators, cytokines and adipocytokines and played an important role in cardiovascular and metabolic disease. Some reports had shown that angiotensin II receptor blockers (ARB) may improve metabolic profiles in patients with diabetes or metabolic syndrome, in addition to its hypotensive effect. It has been reported that some ARB, such as telmisartan and candesartan, can prevent weight gain and high-fat-induced obesity in experimental animals. However, whether telmisartan intervention on improvement of fat deposition and other related metabolic profiles is better than a CCB drugs (amlodipine) in those obese hypertensive patients with diabetes, was still unknown.

ELIGIBILITY:
Inclusion Criteria:

* Information Consent Signed
* Aged 30~70 years
* For whom without anti-hypertensive therapy in 2 weeks：140mmHg≤SBP<180mmHg，或90mmHg≤DBP<110mmHg. For whom with anti-hypertensive therapies in 2 weeks：SBP<180mmHg, 且DBP<110mmHg
* Waist circumference higher than 90cm in men, 80cm in women
* Diagnosed diabetes

Exclusion Criteria:

* Grade 3 hypertension: SBP≥180mmHg, or DBP≥110mmHg
* Waist circumference less than 90cm in men, 80cm in women
* Known allergy or hypersensitivity to trial drugs
* NYHA grade Ⅱ~Ⅳ heart failure, Myocardial infarction or cerebrovascular accident in 1 year preceding the trial
* Acute infections, tumor, severe arrhythmia, mental disease, drug or alcohol abuse
* History of hepatitis or cirrhosis
* History of severe kidney disease
* Pregnant, lactation
* Enrolled in other trials in 3 months
* Any obstacles of follow-up or compliance

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, 24 weeks(End of trial)
Metabolic profiles, including lipid profile and blood glucose | Baseline, 24 weeks(End of trial)

SECONDARY OUTCOMES:
Abdominal fat assessed by CT | Baseline, 24 weeks(End of trial)
Obesity parameters, including waist circumference (WC) and body mass index (BMI) | Baseline, 24 weeks(End of trial)
Incidents of side effects between groups | Baseline, 24 weeks(End of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zhu, MD, PhD, Principal Investigator — The third hospital affiliated to the Third Military Medical University. China
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, China